CLINICAL TRIAL: NCT03466424
Title: Phase I Trial of Dose-escalation Preoperative Short-course Radiotherapy (5×6Gy/7Gy/8Gy) Followed by Neo-adjuvant Chemotherapy in Locally Advanced Rectal Cancer : the FJUHR-01 Trial
Brief Title: Short-course Radiotherapy (5×6Gy/7Gy/8Gy) Followed by Neo-adjuvant Chemotherapy for Locally Advanced Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Benhua Xu, Director,Radiation Oncology, Fujian Medical University Union Hospital
Other Study IDs: FujianUnionH
Record Dates: First submitted 2018-02-28; First posted 2018-03-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Radiation Oncology; Rectal Cancer
Keywords: Short-course radiotherapy; dose escalation; neo-adjuvant chemotherapy; mFOLFOX6; rectal cancer; Phase I trial
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, tumor tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: preoperative short-course radiotherapy(5×6Gy) followed by 4×mFOLFOX6 chemotherapy
  Interventions: Radiation: preoperative short-course radiotherapy
- Group 2: preoperative short-course radiotherapy(5×7Gy) followed by 4×mFOLFOX6 chemotherapy
  Interventions: Radiation: preoperative short-course radiotherapy
- Group 3: preoperative short-course radiotherapy(5×8Gy) followed by 4×mFOLFOX6 chemotherapy
  Interventions: Radiation: preoperative short-course radiotherapy

INTERVENTIONS:
Radiation: preoperative short-course radiotherapy — Patients will be enrolled into Group 1 to 3 according to the time order of entering the study to receive dose from 6Gy×5F to 8Gy×5F using the traditional 3+3 dose escalation design.
  Other Names: 4 cycles mFOLFOX6 chemotherapy

SUMMARY:
Preoperative radiotherapy followed by total mesorectal excision (TME) has been recommended as the preferred treatment method for locally advanced rectal cancer. Similar rates of local control, survival and toxicity were observed in preoperative long-course radiotherapy (LCRT) (45-50.4 Gy in 25-28 fractions) and short-course radiotherapy (SCRT) of 25 Gy in five fractions. For the convenience of SCRT, a growing number of patients tend to receive SCRT as preoperative radiotherapy. Although SCRT can shorten treatment interval and cut down the cost of treatment, it's pathological complete response (pCR) rate is relatively low (SCRT vs. LCRT: 0.7% vs. 16%). Hence, the optimal pattern of preoperative therapy of locally advanced rectal cancer still deserves to be explored. Previous studies have confirmed the feasibility and safety of 30Gy/5 fractions in SCRT of rectal cancer and verified that SCRT followed by mFOLFOX6 chemotherapy can improve the pCR rates. Therefore, investigators aimed to establish a dose escalation mode of SCRT (5×6Gy/7Gy/8Gy) followed by four cycles of modified FOLFOX6(mFOLFOX6) chemotherapy to test the safety and efficacy in treating locally advanced rectal cancer.

DETAILED DESCRIPTION:
Rectal cancer is one of the most common malignant tumors in western countries and its incidence and mortality rates have been ascending for several decades in our country. Surgical resection is the primary treatment method for resectable tumor. Post-operative chemo-radiotherapy can improve local control but can also lower the tolerance rate and increase the incidence of postoperative complications. It is generally not recommended as a regular treatment method excepting the patients who have high risk factors of recurrence after surgery. Preoperative radiotherapy followed by total mesorectal excision(TME) has been recommended as a preferred treatment regimen for locally advanced rectal cancer for it is more effective in local control compared with that of postoperative radiotherapy. The traditional long-course radiotherapy(LCRT) is 45-50.4 Gy in 25-28 daily fractions given with concurrent chemotherapy and delayed surgery(4-8 weeks after chemo-radiotherapy). Also considered an alternative treatment option is preoperative short-course radiotherapy(SCRT) of 25 Gy in five daily fractions and followed by immediate surgery(1 week after SCRT). Similar rates of local control, survival and toxicity were observed in these two regimens. Although SCRT can reduce treatment interval and cut down costs, it's pathological complete response(pCR) rates are relatively low. Bujko et al. reported that the pCR rate for LCRT and SCRT are 16% and 0.7%, respectively. This difference may partially related to the interval between preoperative radiotherapy and surgery. The pCR rates are higher in patients who have the longer interval. In the latest multicenter, randomized, non-blinded, phase III, non-inferiority trial(Stockholm III), participants were randomly assigned to receive either 5×5 Gy radiation dose with immediate surgery within 1 week(SCRT) or after 4-8 weeks(SCRT with delay) or 25×2 Gy radiation dose followed by surgery after 4-8 weeks(LCRT with delay). All these regimens show similar oncological results. However, LCRT with delay prolongs the treatment interval substantially. Although radiation-induced toxicity was observed after SCRT with delay, postoperative complications were significantly reduced compared with that of SCRT followed by immediate surgery. Thus, SCRT with delay to surgery is a useful alternative to conventional SCRT with immediate surgery.

The optimal pattern of dose fractionation of preoperative radiotherapy still deserves to be explored. J Widder et al. reported that SCRT of 25 Gy administered within 1 week of 2.5 Gy twice daily for resectable rectal cancer generates a well-tolerated and simple way to increase local control. A prospective phase II study of SCRT for rectal cancer with twice daily fractions of 2.9 Gy to a total dose of 29 Gy also results in tolerable toxicity and favourable local control. Although both of the modifications of SCRT have acceptable toxicity and well local control, the improvement in overall survival is still limited. Investigators suppose that whether escalating single radiation dose of SCRT (6Gy,7Gy,8Gy...) may further improve local control and overall survival with tolerable toxicity. A prospective phase II study of SCRT that made a boost to the gross tumor volume(GTV) up to a total of 30 Gy in five fractions to investigate the feasibility and the rate of complete pathological response. The results demonstrated that acceptable toxicity and a better rate of pCR can be achieved. Studies have confirmed that high pCR rates were beneficial to survival. Hence, investigators consider that it is feasible to escalate single radiation dose of SCRT in treating rectal cancer. The theoretical basis of escalation of single radiation dose of SCRT may improve survival outcome are as follows:

1. To improve the biological equivalent doses(BED) of the tumor Biological equivalent doses (BED) were used for comparison of various fractionations of radiotherapy and were calculated with the formula for late normal tissue toxicity BED (Gy) =nd[1 +(d /α / β)] n: number of fractions d: single fraction dose (Gy) α/β: take 3 Gy for normal tissues According to the formula, BED is determined by n, d and α/β. This suggests that escalation of fractional dose can significantly increase BED of tumor, thus can amount to the greater kill to tumor cells.
2. To induce tumor immune response Several studies reported that radiotherapy can induce or regulate immune response, which can suppress tumor growth and generate inflammatory response. Field radiotherapy can motivate the radiation effects of local-regional and distant area of the body.

The other one criticism in treating rectal cancer is distant metastasis that hinder the improve of overall survival. Preoperative chemotherapy can play a role in controlling the potential micrometastases. Previous studies have confirmed that SCRT followed by mFOLFOX6 chemotherapy can improve the pCR rates. Therefore, in this Phase I Study, the safety and efficacy will be tested using a dose escalation mode of SCRT (5×6Gy/7Gy/8Gy) followed by four cycles of mFOLFOX6 chemotherapy when treating locally advanced rectal cancer.

Dose Escalation Methods in Phase I Cancer Clinical Trials:

Three patients receive the lowest level of radiation dose in a cohort and dose limited toxicity(DLT) is observed. If none of the patients show DLT, another cohort of three patients receive the next higher level of dose. If not, a further cohort of three patients will receive the same dose when one or more patients exhibit DLT. Of the six patients treated at this dose level, the trial continues at the next dose level if only one out the six patients appears DLT and stops at that dose level if at least two patients appear DLT. When the escalation stopped, additional three patients will be required at this dose level. The maximum sample size will depend on the dose level that is in progress.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated, biopsy-proven stage T3-4 and/or N+，resectable rectal adenocarcinoma with the tumors near anal verge within 12 cm;
* Male or non-pregnant female;
* Between 18 and 70 years of age;
* Adequate hematologic function: white blood cell(WBC) counts≥4,000/mm3, neutrophils counts ≥ 1,500/mm3, platelet counts ≥ 100,000/µL, hemoglobin ≥ 9g/L;
* Adequate renal function: creatinine ≤ 1.5×upper normal limit;
* Adequate hepatic function: total bilirubin, glutamic oxalacetic transaminase, glutamate pyruvate transaminase level < 2.0×upper normal limit);
* Satisfactory performance status: Karnofsky Performance Status(KPS)≥70;
* Approval from the ethics committee and prior written informed consents from all patients before registration were obtained.

Exclusion Criteria:

* the evidence of relapse or distant metastasis;
* receiving treatment of other anti-cancer drugs or methods;
* Patients have low compliance and are not able to complete the entire trial;
* the presence of uncontrolled life-threatening diseases;
* dysfunction of heart, brain, lung and et al.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hosptal in-patients
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response(pCR) rate | four weeks after surgery
  According to pathological response criteria, a total regression is considered a complete response.

SECONDARY OUTCOMES:
R0 resection rate | four weeks after surgery
  According to the pathological outcomes after received surgery.
Sphincter preservation rate | four weeks after surgery
  According to the pathological outcomes after received surgery.
Incidence of surgical complications | four weeks after surgery
  Surgical complications are defined as those occurring within 30 days after surgery, such as re-operation, anastomotic fistula, bleeding, infection and death related to the operation.
Incidence of acute toxicities during radiation or chemotherapy | three months
  Number of participants with abnormal laboratory values and/or adverse events that are related to radiation or chemotherapy as assessed by Common Toxicity Criteria for Adverse Effects(CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Benhua Xu, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Zhang MX, Li XB, Guan BJ, Guan GX, Lin XY, Wu XD, Chi P, Xu BH. Dose escalation of preoperative short-course radiotherapy followed by neoadjuvant chemotherapy in locally advanced rectal cancer: protocol for an open-label, single-centre, phase I clinical trial. BMJ Open. 2019 Mar 23;9(3):e025944. doi: 10.1136/bmjopen-2018-025944. PMID 30904869